CLINICAL TRIAL: NCT00095979
Title: A Phase II Evaluation of Ixabepilone (BMS-247550) [NCI-Supplied Agent, NSC #710428]) in the Treatment of Recurrent or Persistent Endometrial Carcinoma
Brief Title: Ixabepilone in Treating Patients With Recurrent or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Gynecologic Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02628; NCI-2012-02628 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000391849; GOG-0129P (Other: Gynecologic Oncology Group); GOG-0129P (Other: CTEP); U10CA027469 (NIH)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Endometrial Adenocarcinoma; Recurrent Endometrial Carcinoma; Stage IV Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — ixabepilone

ARMS (1):
- Treatment (ixabepilone) (Experimental): Patients receive ixabepilone IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: ixabepilone

INTERVENTIONS:
Drug: ixabepilone — Given IV
  Other Names: BMS-247550; epothilone B lactam; Ixempra

SUMMARY:
Drugs used in chemotherapy, such as ixabepilone, work in different ways to stop tumor cells from dividing so they stop growing or die. This phase II trial is studying how well ixabepilone works in treating patients with recurrent or persistent endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate in patients with recurrent or persistent endometrial adenocarcinoma treated with ixabepilone.

II. Determine the nature and degree of toxicity of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive ixabepilone IV over 3 hours on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: A total of 19-51 patients will be accrued for this study within 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial adenocarcinoma

  * Recurrent or persistent disease

    * Histologic confirmation of the original primary tumor is required
  * Not amenable to management with any of the following:

    * Surgery
    * Radiotherapy
    * Higher priority or standard chemotherapy
* Measurable disease

  * At least 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques (e.g., palpation, plain x-ray, CT scan, or MRI) OR ≥ 10 mm by spiral CT scan
* At least 1 target lesion

  * Tumors within a previously irradiated field are designated as non-target lesions
  * Disease in an irradiated field as the only site of measurable disease is acceptable as a target lesion only if there has been clear progression of the lesion at least 90 days after completion of radiotherapy
* Received 1, and only 1, prior chemotherapy regimen (e.g., high-dose therapy, consolidation, or extended therapy administered after surgery or non-surgical assessment) for management of endometrial adenocarcinoma
* Ineligible for a higher priority Gynecologic Oncology Group (GOG) protocol (e.g., any active GOG phase III study for the same patient population)
* Performance status - GOG 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST (aspartate aminotransferase) ≤ 2.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Sensory or motor neuropathy ≤ grade 1
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection requiring antibiotics
* No other invasive malignancies within the past 5 years except non-melanoma skin cancer
* At least 3 weeks since prior biologic or immunologic agents directed at the malignant tumor
* One prior non-cytotoxic* (biologic or cytostatic) regimen for management of recurrent or persistent disease allowed
* See Disease Characteristics
* Prior paclitaxel or docetaxel allowed
* Recovered from prior chemotherapy
* No more than 1 prior cytotoxic chemotherapy regimen (either single or combination drug therapy)
* No prior ixabepilone
* At least 1 week since prior hormonal therapy directed at the malignant tumor

  * Continuation of hormone replacement therapy allowed
* See Disease Characteristics
* Recovered from prior radiotherapy
* Recovered from prior surgery
* At least 3 weeks since other prior therapy directed at the malignant tumor
* No prior cancer treatment that contraindicates study therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2005-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Dizon, Principal Investigator — Gynecologic Oncology Group
Locations (1):
- Gynecologic Oncology Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 5/2/2005 and closed to accrual on 1/3/2008 (suspended from 4/3/2006 to 4/1/2007).
Groups:
- Ixabepilone: Ixabepilone 40 mg/m2 administered as 3-hour infusion on day 1 of a 21-day cycle until disease progression or adverse effects prohibit further treatment
Period: Overall Study
Arm/Group | Ixabepilone
Started | 52
Completed | 50
Not Completed | 2
Not completed — Ineligible: Second primary cancer site | 2

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients
Arm/Group | Ixabepilone
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.8 (9.4)
Age, Customized [Number; unit: participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 2
  50-59 years | 11
  60-69 years | 19
  70-79 years | 16
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
International Federation of Gynecology and Obstetrics (FIGO) Stage Recurrent/Persistent [Number; unit: participants] | 50
Histologic Type [Number; unit: participants]
  Adenocarcinoma, Unspecified | 1
  Clear Cell Carcinoma | 1
  Endometrioid Adenocarcinoma | 22
  Mixed Epithelial Carcinoma | 4
  Serous Adenocarcinoma | 21
  Carcinosarcoma-homologous | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: RECIST 1.0 defines complete response as the disappearance of all target lesions and non-target lesions and no evidence of new lesions documented by two disease assessments at least 4 weeks apart. Partial response is defined as at least a 30% decrease in the sum of longest dimensions (LD) of all target measurable lesions taking as reference the baseline sum of LD. There can be no unequivocal progression of non-target lesions and no new lesions. Documentation by two disease assessments at least 4 weeks apart is required. In the case where the ONLY target lesion is a solitary pelvic mass measured by physical exam, which is not radiographically measurable, a 50% decrease in the LD is required. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: Every other cycle for first 6 months; then every six months thereafter until completion of study treatment; and at any other time if clinically indicated based on symptoms or physical signs suggestive of progressive disease
Population: Eligible and Treated Patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Ixabepilone
Number analyzed (Participants) | 50
percentage of participants | 12 [7 to 100]

2. Primary Outcome: Frequency and Severity of Observed Adverse Effects Associated With Protocol Therapy (CTCAE Version 3)
Time Frame: Every cycle until completion of study treatment up to 30 days after stopping study treatment (average length of data collection = 4 months)
Population: Eligible and treated patients
Measure: Count of Participants; unit: Participants
Groups:
- Grade 1: Number of patients who experienced a grade 1 event using Common Terminology Criteria for Adverse Events (CTCAE version 3).
- Grade 2: Number of patients who experienced a grade 2 event using Common Terminology Criteria for Adverse Events (CTCAE version 3).
- Grade 3: Number of patients who experienced a grade 3 event using Common Terminology Criteria for Adverse Events (CTCAE version 3).
- Grade 4: Number of patients who experienced a grade 4 event using Common Terminology Criteria for Adverse Events (CTCAE version 3).
- Grade 5: Number of patients who experienced a grade 5 event using Common Terminology Criteria for Adverse Events (CTCAE version 3).
Arm/Group | Grade 1 | Grade 2 | Grade 3 | Grade 4 | Grade 5
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 50
Participants
  Leukopenia | 9 | 14 | 17 | 7 | 0
  Neutropenia | 5 | 7 | 14 | 12 | 0
  Anemia | 12 | 29 | 6 | 1 | 0
  Thrombocytopenia | 13 | 4 | 1 | 1 | 0
  Allergy/Immunology | 4 | 0 | 0 | 0 | 0
  Auditory/ear | 0 | 2 | 0 | 0 | 0
  Cardiac | 1 | 0 | 2 | 0 | 0
  Coagulation | 0 | 0 | 1 | 0 | 0
  Constitutional | 15 | 14 | 9 | 1 | 0
  Dermatologic | 7 | 21 | 2 | 0 | 0
  Gastrointestinal | 11 | 15 | 12 | 0 | 0
  Genitourinary | 1 | 1 | 0 | 0 | 0
  Hemorrhage | 1 | 1 | 2 | 0 | 0
  Infection | 0 | 2 | 8 | 0 | 0
  Lymphatics | 8 | 2 | 0 | 0 | 0
  Metabolic | 9 | 8 | 3 | 1 | 0
  Musculoskeletal | 3 | 4 | 0 | 0 | 0
  Neurosensory | 19 | 7 | 4 | 0 | 0
  Other neurologic | 4 | 3 | 4 | 1 | 0
  Ocular/visual | 3 | 3 | 0 | 0 | 0
  Pain | 9 | 8 | 3 | 0 | 0
  Pulmonary | 10 | 4 | 2 | 0 | 1
  Alopecia | 7 | 23 | 0 | 0 | 0
  Vascular | 0 | 1 | 0 | 1 | 0

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined according to RECIST v1.0 as at least a 20% increase in the sum of LD target lesions taking as reference the smallest sum LD recorded since study entry, the appearance of one or more new lesions, death due to disease without prior objective documentation of progression, global deterioration in health status attributable to the disease requiring a change in therapy without objective evidence of progression, or unequivocal progression of existing non-target lesions.
Time Frame: From study entry to disease progression, death or date of last contact, whichever occurs first, up to 5 years of follow-up.
Population: Eligible and Treated Patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone
Number analyzed (Participants) | 50
months | 3.1 [2.8 to 4.2]

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: From study entry to death or last contact, up to 5 years of follow-up.
Population: Eligible and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ixabepilone
Number analyzed (Participants) | 50
months | 8.8 [6.3 to 11.9]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported. Average length of data collection = 4 months.
Arm/Group | Ixabepilone
Serious Adverse Events (participants affected / at risk) | 25/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=50)
Neutrophils (Blood and lymphatic system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 1
S/N Arrhythmia: Atrial Fibrillation (Cardiac disorders) | 1
Fatigue (General disorders) | 1
Death No Ctcae Term - Disease Progression Nos (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1
Febrile Neutropenia (Infections and infestations) | 2
Creatinine (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Syncope (Nervous system disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 2
Pain: Tumor (General disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone (N=50)
Allergic Reaction/Hypersensitivity (Immune system disorders) | 2
Rhinitis (Immune system disorders) | 4
Hearing (Without Monitoring Program) (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Neutrophils (Blood and lymphatic system disorders) | 36
Platelets (Blood and lymphatic system disorders) | 20
Leukocytes (Blood and lymphatic system disorders) | 47
Lymphopenia (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 48
Supraventricular Tachycardia (Cardiac disorders) | 1
Ventricular Arrhythmia - Pvcs (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Hypotension (Cardiac disorders) | 3
Inr (Vascular disorders) | 1
Sweating (General disorders) | 3
Patient Odor (General disorders) | 1
Fever (General disorders) | 5
Weight Loss (General disorders) | 4
Rigors/Chills (General disorders) | 4
Fatigue (General disorders) | 40
Insomnia (General disorders) | 7
Nail Changes (Skin and subcutaneous tissue disorders) | 6
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 30
Bruising (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Flushing (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
Hot Flashes (Endocrine disorders) | 1
Diabetes (Endocrine disorders) | 1
Hypoparathyroidism (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Heartburn (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Leak, Gi - Rectum (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Taste Alteration (Gastrointestinal disorders) | 6
Dry Mouth (Gastrointestinal disorders) | 1
Mucositis (Functional/Sympt) - Oral Cavity (Gastrointestinal disorders) | 4
Obstruction, Gi - Small Bowel Nos (Gastrointestinal disorders) | 1
Mucositis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 6
Mucositis (Clinical Exam) - Esophagus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 19
Anorexia (Gastrointestinal disorders) | 25
Dehydration (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 24
Nausea (Gastrointestinal disorders) | 22
Diarrhea (Gastrointestinal disorders) | 22
Hemorrhage, Gu - Urinary Nos (Vascular disorders) | 2
Hemorrhage, Gu - Vagina (Vascular disorders) | 4
Hemorrhage, Gi - Rectum (Vascular disorders) | 2
Hemorrhage, Gi - Upper Gi Nos (Vascular disorders) | 1
Hemorrhage/Pulmonary - Nose (Vascular disorders) | 2
Hemorrhage, Gu - Bladder (Vascular disorders) | 1
Inf W/Gr 3 Or 4 Anc: Blood (Infections and infestations) | 1
Inf W/Gr 3 Or 4 Anc: Middle Ear (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Oral Cavity-Gums (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Catheter-Related (Infections and infestations) | 1
Febrile Neutropenia (Infections and infestations) | 3
Inf W/Nml Or Gr 1 Or 2 Anc: Urinary Tract Nos (Infections and infestations) | 1
Infection - Other (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Conjunctiva (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bronchus (Infections and infestations) | 1
Inf Unknown Anc: Urinary Tract Nos (Infections and infestations) | 7
Inf Unknown Anc: Bladder (Urinary) (Infections and infestations) | 1
Inf Unknown Anc: Lip/Perioral (Infections and infestations) | 1
Inf W/Gr 3 Or 4 Anc: Upper Airway Nos (Infections and infestations) | 1
Inf W/Nml Or Gr 1 Or 2 Anc: Bladder (Infections and infestations) | 2
Inf W/Gr 3 Or 4 Anc: Urinary Tract Nos (Infections and infestations) | 4
Edema: Limb (Blood and lymphatic system disorders) | 12
Ast (Metabolism and nutrition disorders) | 4
Gfr (Metabolism and nutrition disorders) | 1
Proteinuria (Metabolism and nutrition disorders) | 3
Hemoglobinuria (Metabolism and nutrition disorders) | 1
Creatinine (Metabolism and nutrition disorders) | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 10
Alt (Metabolism and nutrition disorders) | 1
Alkaline Phosphatase (Metabolism and nutrition disorders) | 4
Bilirubin (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 13
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 14
Hypokalemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 15
Joint-Function (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Whole Body/Generalized (Musculoskeletal and connective tissue disorders) | 3
Muscle Weakness - Left-Sided (Musculoskeletal and connective tissue disorders) | 1
Muscle Weakness - Extremity-Lower (Musculoskeletal and connective tissue disorders) | 2
Mood Alteration - Depression (Nervous system disorders) | 5
Mood Alteration - Anxiety (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 6
Neuropathy-Sensory (Nervous system disorders) | 32
Neuropathy-Motor (Nervous system disorders) | 5
Ocular/Visual - Other (Eye disorders) | 2
Uveitis (Eye disorders) | 1
Watery Eye (Eye disorders) | 2
Dry Eye (Eye disorders) | 1
Flashing Lights/Floaters (Eye disorders) | 1
Blurred Vision (Eye disorders) | 5
Eyelid Dysfunction (Eye disorders) | 1
Pain: Pelvis (General disorders) | 2
Pain: Breast (General disorders) | 1
Pain: Vagina (General disorders) | 1
Pain: Chest /Thorax Nos (General disorders) | 3
Pain: Chest Wall (General disorders) | 1
Pain: Eye (General disorders) | 1
Pain: Head/Headache (General disorders) | 7
Pain: Extremity-Limb (General disorders) | 11
Pain: Back (General disorders) | 8
Pain: Joint (General disorders) | 6
Pain: Bone (General disorders) | 3
Pain: Kidney (General disorders) | 1
Pain: Bladder (General disorders) | 2
Pain: Pain Nos (General disorders) | 2
Pain: Stomach (General disorders) | 2
Pain: Oral Cavity (General disorders) | 1
Pain: Abdominal Pain Nos (General disorders) | 14
Pain: Middle Ear (General disorders) | 1
Pain: Tumor (General disorders) | 1
Pain: Muscle (General disorders) | 8
Pain: Neuralgia (General disorders) | 2
Voice Changes (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Leak, Gu - Vagina (Renal and urinary disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Urinary Retention (Renal and urinary disorders) | 1
Obstruction, Gu - Ureter (Renal and urinary disorders) | 1
Incontinence, Urinary (Renal and urinary disorders) | 4
Bladder Spasm (Renal and urinary disorders) | 1
Urinary Frequency (Renal and urinary disorders) | 2
Vaginal Discharge (Reproductive system and breast disorders) | 1
Thrombosis/Thrombus/Embolism (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less